CLINICAL TRIAL: NCT02790307
Title: Single Centre Randomised Pilot Study of Two Regimens (30mins Daily or Weekly for 12 Weeks) of Transcutaneous Tibial Nerve Stimulation of Patients With Overactive Bladder (OAB) Syndrome
Brief Title: Transcutaneous Tibial Nerve Stimulation of Patients With Overactive Bladder (OAB) Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Jalesh Panicker, Consultant Uro-Neurologist and Honorary Senior Lecturer, University College, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/LO/1613
Record Dates: First submitted 2016-04-07; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Overactive Bladder; Multiple Sclerosis
Keywords: multiple sclerosis; overactive bladder; urinary incontinence; tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Multiple Sclerosis; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily stimulation (30mins/day) (Experimental): 30 minutes daily for 12 weeks of Tibial nerve stimulation using the Geko device
  Interventions: Device: The Geko
- Weekly stimulation (30mins/week) (Experimental): 30 minutes daily for 12 weeks of Tibial nerve stimulation using the Geko device
  Interventions: Device: The Geko

INTERVENTIONS:
Device: The Geko — transcutaneous tibial nerve stimulation (stick on patch)

SUMMARY:
Tibial nerve stimulation (TNS) has been recognised as a safe and effective treatment for the management of overactive bladder (OAB) symptoms. The aim of this study was to evaluate safety, acceptability and pilot efficacy of transcutaneous TNS using a novel device.

DETAILED DESCRIPTION:
In this single centre pilot study, 48 patients with OAB (24 with neurogenic and 24 with idiopathic OAB) were randomized to use a self-applicating ambulatory skin-adhering device to transcutaneously stimulate the tibial nerve for 30 minutes, either once daily or once weekly, for 12-weeks. Changes in lower urinary tract (LUT) OAB symptoms and QoL were measured at baseline, weeks 4, 8, and 12 using standardized validated scoring instruments (ICIQ-OAB and ICIQ-LUTSqol) and a Global Response Assessment (GRA) at week 12. Weekly phone calls and a usage diary captured patient-reported experiences with the device and compliance.

The primary study outcomes were to assess safety and acceptability of the device. In addition, treatment response was assessed using the Global Response Assessment (GRA) at week-12, and the International Consultation on Incontinence Questionnaire Overactive Bladder and LUTS-quality of life (ICIQ-OAB and ICIQ-LUTSqol) at baseline, week 4, 8 and 12. In the GRA patients were asked to assess their response to treatment using an ordinal scale of 0 to 3, referring to none, mild, moderate or marked improvement, respectively 1. Patients reporting moderate or marked improvement were considered to have responded to treatment 1. The ICIQ-OAB score is a 4-item questionnaire that assesses OAB symptom severity and bother whereas the ICIQ-LUTSqol score is a 20-item health related quality of life questionnaire. In both questionnaires, part A assesses symptom severity and part B reflects the accumulative bother to the patient. High scores suggests worse symptom profiles and negative impact on QoL, respectively.

Patients recorded use of the device in a customized compliance diary which also included entries for their experiences in using the device and any adverse effects. Additionally, weekly phone calls were made by a member of the research team to assess compliance.

Statistical analysis A feasibility sample size of 48 patients was adopted and no formal power calculation was performed as is the convention for pilot studies. All data were presented as means with SDs. Paired student t-tests were used to provide an estimate of within group responses between baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility was based on meeting the criteria for an overactive bladder, defined by the International Continence Society with an average urinary frequency ≥ 8 voids per and ≥ 1 urgency episode (with or without incontinence) per 24 hours

Exclusion Criteria:

* Exclusion criteria included use of botulinum toxin A treatment within the previous year or neuromodulation (TNS or sacral neuromodulation), patients with sensory loss in the gaitor region (based on intact cutaneous sensation to nociception in the lower limb), presence of urinary tract infection or any other documented LUT pathology

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting adverse events as recorded using a customised diary | 12 weeks
  Adverse events are recorded by patients using a compliance diary

SECONDARY OUTCOMES:
Improvement in overactive bladder symptoms as evaluated using a Global Response Assessment (GRA) scale | 12 weeks
  The Global Response Assessment (GRA) scale assesses the response to treatment using an ordinal scale of 0 to 3, referring to none, mild, moderate or marked improvement, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jalesh Panicker, FRCP, Principal Investigator — National Hospital for Neurology and Neurosurgery
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] de Seze M, Raibaut P, Gallien P, Even-Schneider A, Denys P, Bonniaud V, Game X, Amarenco G. Transcutaneous posterior tibial nerve stimulation for treatment of the overactive bladder syndrome in multiple sclerosis: results of a multicenter prospective study. Neurourol Urodyn. 2011 Mar;30(3):306-11. doi: 10.1002/nau.20958. Epub 2011 Feb 8. PMID 21305588